CLINICAL TRIAL: NCT04232410
Title: Measurement of Critical Closing Pressure (Pcrit) During Drug-Induced Sleep Endoscopy (DISE)
Acronym: Pcrit-DISE
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, Prof. Dr. Olivier Vanderveken, University Hospital, Antwerp
Other Study IDs: BE300201940940
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSA Pcrit-DISE: Patients diagnosed with OSA and eligible for non-CPAP treatments
  Interventions: Diagnostic Test: Drug induced sleep endoscopy; Diagnostic Test: Measurement of critical closing pressure of the uppper airway

INTERVENTIONS:
Diagnostic Test: Drug induced sleep endoscopy — DISE is performed in a semi-dark, silent operating theatre, starting with the patient in supine position. To first induce sleep, an IV bolus of midazolam (1.5 mg) is administered. Then, a flexible fiberoptic nasopharyngoscope (Olympus END-GP, 3.7 mm diameter, Olympus Europe GmbH, Hamburg, Germany) is inserted through one of the nostrils. Either at the start of the examination or while holding the scope at the level of the palate, propofol (2.0-3.0 µg/ml) will be administered via a target-controlled infusion (TCI) pump. Sleep occurrence is confirmed using the additional EEG measurement.
  Other Names: DISE
Diagnostic Test: Measurement of critical closing pressure of the uppper airway — After sleep onset, the CPAP pressure well be increased until no flow limitations are observed. This pressure is called the holding pressure and is used as a base for all the following measurements for that individual OSA patient. After observing sleep stage 2 or 3, the holding pressure is reduced abruptly by 1 cmH2O during expiration for 5 breaths. Then the pressure is set back to the holding pressure for the duration of 1 minute. This procedure is repeated until obstructive sleep apnea is noted.
  Other Names: Pcrit measurement

SUMMARY:
This study intends to test the feasibility of measurement of the critical closing pressure (Pcrit) during drug-induced sleep endoscopy (DISE) for use in future studies, which are aimed at finding an alternative method for patient selection and response prediction before implementation of non-CPAP therapies.Twenty patients diagnosed with OSA and eligible for non-CPAP treatments are going to be included into this study and undergo these measurements. Drug-induced sleep endoscopy (DISE) is part of the standard clinical care for OSA patients that are eligible for non-CPAP therapies. We aim to expand this procedure with measurement of Pcrit, oesophageal pressure, airflow, EEG, EOG, respiratory effort, SpO2 and chin EMG during this study.

DETAILED DESCRIPTION:
Patients from the ENT department will be recruited and informed about the study. After obtaining informed consent, the patients will undergo DISE according to the normal clinical care.The study will be performed during this clinical DISE, using a standard polysomnographic set-up (Alice 6 LDx, Philips Respironics) expanded with pressure and flow measurements. After measurements and evaluations are done, the most suitable treatment option based on the DISE and PSG findings, as defined in the standard clinical care, will be advised to the patient. The treatment and its further choice are not part of the current study protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis with OSA (AHI ≥15/hour sleep)
* Eligible for DISE as the next step in the clinical path for OSA.
* Capable of giving informed consent

Exclusion Criteria:

* Medication use related to sleeping disorders.
* Central sleep apnea syndrome.
* Medical history of known causes of tiredness or severe sleep disruption other than OSA (insomnia, PLMS, Narcolepsy).
* Seizure disorder.
* Known medical history of intellectual disability, memory disorders or current psychiatric disorders (psychotic illness, major depression, or acute anxiety attacks as mentioned by the patient).
* Inability to provide informed consent.
* Simultaneous use of other treatment modalities to treat OSA
* Esophageal ulceration, tumors, diverticulitis, bleeding varices, sinusitis, epistaxis, recent nasopharyngeal surgery
* Pregnancy or willing to become pregnant
* Excessive alcohol or drug use (> 20 alcohol units/week or any use of hard drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty patients diagnosed with OSA and eligible for non-CPAP
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Critical closing pressure of the upper airway (Pcrit) | 1 hour
  The pressure at which the upper airway collpases measured in cm H2O.

SECONDARY OUTCOMES:
Airflow | 1 hour
  By using a pneumotachometer attached to a transducer the inspiratory and expiratory airflow (l/s) will be measured.
EEG | 1 hour
  Using electroencephalogram electrodes C3, C4, O1, F4 to evaluate sleep and wake stages and ground and system reference electrodes (volt)
Esophageal pressure | 1 hour
  The pressure of the esophagus measured in cmH2O using an esophageal ballooon catheter.
SpO2 | 1 hour
  using a pulse oximetry device, to non-invasively measure arterial oxygen saturation level (%).
EMG | 1 hour
  Using electromyogram electrodes to evaluate muscular activity (volt)
EOG | 1 hour
  electrooculogram electrodes to evaluate rapid eye movements (volt)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Vanderveken, MD, PhD, Study Chair — Head of ENT department, UZA
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
The patient data is coded and only the investigators will have access to the data.

REFERENCES:
- [Background] Azarbarzin A, Sands SA, Taranto-Montemurro L, Oliveira Marques MD, Genta PR, Edwards BA, Butler J, White DP, Wellman A. Estimation of Pharyngeal Collapsibility During Sleep by Peak Inspiratory Airflow. Sleep. 2017 Jan 1;40(1):zsw005. doi: 10.1093/sleep/zsw005. PMID 28364460
- [Background] Gold AR, Schwartz AR. The pharyngeal critical pressure. The whys and hows of using nasal continuous positive airway pressure diagnostically. Chest. 1996 Oct;110(4):1077-88. doi: 10.1378/chest.110.4.1077. No abstract available. PMID 8874271
- [Derived] Van de Perck E, Kazemeini E, Van den Bossche K, Willemen M, Verbraecken J, Vanderveken OM, Op de Beeck S. The effect of CPAP on the upper airway and ventilatory flow in patients with obstructive sleep apnea. Respir Res. 2023 May 31;24(1):143. doi: 10.1186/s12931-023-02452-z. PMID 37259138
- [Derived] Kazemeini E, Van de Perck E, Dieltjens M, Willemen M, Verbraecken J, Sands SA, Vanderveken OM, Op de Beeck S. Critical closing pressure of the pharyngeal airway during routine drug-induced sleep endoscopy: feasibility and protocol. J Appl Physiol (1985). 2022 Apr 1;132(4):925-937. doi: 10.1152/japplphysiol.00624.2021. Epub 2022 Feb 3. PMID 35112928